CLINICAL TRIAL: NCT04129177
Title: Reduction of Surgical Site Infections in Elective Colorectal Surgery After the Implementation of a Bundle of Preventative Measures. Multicenter Study of the Nococomial Infection Surveillance Program in Catalonia.
Brief Title: Reduction of Surgical Site Infections in Elective Colorectal Surgery After the Implementation of a Bundle of Care.
Status: Completed | Type: Observational
Sponsor: Hospital de Granollers (Other)
Responsible Party: Principal Investigator, Josep M Badia, Director of surgical infection department, Hospital de Granollers
Other Study IDs: HGranollers
Record Dates: First submitted 2019-10-15; First posted 2019-10-16 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Colorectal Neoplasms; Surgical Wound Infection
Keywords: Surgical site infection; Colorectal surgery; Surveillance; Bundle approach
MeSH Terms: conditions — Colorectal Neoplasms; Surgical Wound Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Implementation of a bundle of surgical infection preventive measures — A bundle of six preventative measures is recommended to the VINCat hospitals. Bundle measures were: systemic and oral antibiotic prophylaxis, mechanical bowel preparation (MBP), laparoscopic surgery, maintenance of normothermia, and the use of a double-ring wound retractor.

SUMMARY:
Background. The Nosocomial Infection Surveillance Program in Catalonia (VINCat) monitors SSI in elective colorectal surgery since 2007 in 56 hospitals (7.5 million population). These hospitals perform active and prospective standardized surveillance of elective colorectal resections. Post-discharge surveillance is mandatory up to 30 days after surgery. Between 2007 and 2015, the SSI rate did not change significantly, with a cumulated incidence of 5,491 SSI in a total of 29,006 interventions (19%). In 2015, a working group of VINCat specialists and surgeons from the Catalan Society of Surgery was set up to formulate a specific bundle of SSI preventative measures for colorectal surgery.

Aim. To analyse the effect of a specific bundle for SSI prevention in elective colorectal surgery.

Methods. In 2016, a bundle of six preventative measures was recommended to the VINCat hospitals. Bundle measures were: systemic and oral antibiotic prophylaxis, mechanical bowel preparation (MBP), laparoscopic surgery, maintenance of normothermia, and the use of a double-ring wound retractor. The results of SSI before and after the implementation of the bundle are compared. The results are analysed using the chi-square test (statistical significance p <0.05).

DETAILED DESCRIPTION:
Surgical location infection (ILQ) is the most frequent complication of surgery and an important source of clinical and economic problems for health systems. The reduction of its incidence is important because of its impact on patient comfort and the health resources used. The ILQ includes the categories of: superficial incisional (IIS, affects skin and subcutaneous tissue); deep incisional (IIP, affects deep soft tissues), and organ-space or organ-cavitary (IOE, affects any anatomical structure other than the incision manipulated during the intervention). Surgical procedures are distributed in the categories of clean, clean-contaminated, contaminated and dirty or infected surgery depending on your risk of ILQ.

Elective colorectal surgery belongs to the clean-contaminated surgery category, it is one of the most frequent surgical procedures in Western society and the one with the highest rate of postoperative infection. The ILQ after colorectal procedures represents a measurable indicator of the quality of a health system. Endogenous factors of the patient and exogenous factors related to the surgical procedure are involved in the development of the ILQ.

Despite the introduction of laparoscopy and the standardization of perioperative measures of prophylaxis, the clean-contaminated nature of these procedures, the increase in comorbidities and age of patients and the increase in the complexity of surgical procedures do not improve the Postoperative ILQ rates. It is necessary to investigate the usefulness of complementary prophylactic measures that allow lowering the level of wound contamination and reducing the rate of ILQ.

The grouping of ILQ prevention measures into bundles or packages of measures with a high level of evidence is a strategy that has proven effective in various types of surgical procedures. The overall effectiveness of a package of measures depends on the degree of individual effectiveness of each of the measures included in the bundle.

The Nosocomial Infection Surveillance Program in Catalonia (VINCat) has been monitoring ILQ rates in elective colorectal surgery since 2007 in 55 hospitals. These hospitals perform active and prospective standardized surveillance of elective colorectal resections. Post-discharge surveillance is mandatory up to 30 days after surgery. Between 2007 and 2015, the rate of ILQ did not change significantly, with a cumulative incidence of 5,491 ILQ in a total of 29,006 interventions (19%). Given the persistence of these infection rates, in 2015, an interdisciplinary working group was formed that included infection control nurses, infectious disease specialists, anesthetists and surgeons of the Catalan Society of Surgery. Its objective was to design a specific package of ILQ preventive measures for elective colorectal surgery that could affect the incisional infection and organ / space.

In 2016, a package of 6 measures of prevention of ILQ in colorectal surgery was implanted in hospitals belonging to VINCat.

Ambit. A multicenter study is proposed in 55 hospitals in Catalonia. This is a cohort study of the prospective VINCat database, which collects data on surgical patients with the purpose of improving quality. Sixty-five VINCat hospitals participate in the surveillance of ILQ in colorectal surgery, an effort focused on improving the ILQ in colon and rectal operations since 2007. There are more than 43,000 case records since that date. VINCat hospitals are predominantly public hospitals.

Workgroup. The working group is multicentre and interdisciplinary, including doctors and nurses of different specialties related to the prevention and control of surgical infection (surgical nursing, anesthesia, infectious diseases, infection spread and surgery) of different hospitals in the territory. The working group has a long experience in the surveillance and prevention of nosocomial and surgical infection and with the necessary means to carry out the project.

Recipients The study recipients are all patients undergoing elective colorectal surgery, one of the most frequent major abdominal surgical procedures in our hospitals and one of the ones that causes the most complications and health costs.

Hypothesis. Implantation of a package of ILQ prevention measures in colorectal surgery, which includes the combination of oral antibiotic and mechanical colon preparation (PMC) may decrease the rate of ILQ in elective colon surgery.

Goals. Principal. Evaluate the effect of the implementation of a package of specific measures (bundle) in reducing the ILQ rate

ELIGIBILITY:
Inclusion Criteria:

* Elective colorectal resection

Exclusion Criteria:

* Emergency surgery - Infection present at operation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing elective colorectal surgery in Catalonia in the period 2012-2018
Sampling Method: Non-Probability Sample
Enrollment: 12000 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Surgical site infection rate | 30 days
  Rate of Surgical site infection according to the definitions of the CDC-NHSN (Centers for Disease Control and Prevention-National Healthcare Safety Network)

CONTACTS AND LOCATIONS:
Locations (1):
- Fundació Privada Hospital Asil de Granollers, Granollers, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Badia JM, Arroyo-Garcia N, Vazquez A, Almendral A, Gomila-Grange A, Fraccalvieri D, Pares D, Abad-Torrent A, Pascual M, Solis-Pena A, Puig-Asensio M, Pera M, Gudiol F, Limon E, Pujol M; Members of the VINCat Colorectal Surveillance Team; VINCat Program*. Leveraging a nationwide infection surveillance program to implement a colorectal surgical site infection reduction bundle: a pragmatic, prospective, and multicenter cohort study. Int J Surg. 2023 Apr 1;109(4):737-751. doi: 10.1097/JS9.0000000000000277. PMID 36917127